CLINICAL TRIAL: NCT05162183
Title: Replication of the LEAD-2 Diabetes Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-LEAD2
Record Dates: First submitted 2021-09-20; First posted 2021-12-17 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — glimepiride; Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Glimepiride: Reference Group
  Interventions: Drug: Glimepiride
- Liraglutide: Exposure group
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Glimepiride — Glimepiride dispensing claim is used as the reference group.
  Groups: Glimepiride
Drug: Liraglutide — Liraglutide dispensing claim is used as the exposure group.
  Groups: Liraglutide

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates through standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes mellitus [0,0] days
* 3 or more recorded HbA1c values [-365, 0] days
* At least two dispensing claims for metformin [-180,0] days
* 1 or more recorded HbA1c values [-90,0] days
* Age between 18-80 [0,0] days

Exclusion Criteria:

* Cancer, malignant neoplasm, or MEN2 [-1,825,0] days
* Use of other anti-diabetic medications [-180,0] days
* Cirrhosis or Hepatic decompensation [-180,0] days
* Viral hepatitis B or C [-180,0] days
* Stage 5 CKD, ESRD, dialysis or renal transplant [-180,0] days
* MI or HF [-180,0] days
* Treatment with Anti-VEGFi or Photocoagulation [-180,0] days
* Hypertensive crisis or uncontrolled hypertension [-180,0] days
* Two diagnoses of hypoglycemia [-180,0] days
* Alcohol/drug abuse/dependence [-180,0] days
* Dementia and brain damages or non-compliance [-180,0] days
* Pregnancy [-180,0] days
* Type 1 DM, DKA, or other metabolic acidosis [-180,0] days
* Systemic corticosteroids [-90,0] days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, propensity score-matched, retrospective cohort design comparing injectable subcutaneous liraglutide (1.2 or 1.8 mg/day) to oral glimepiride (4 mg once daily). Treatments in both arms are administered in combination with metformin (up to 2,000 mg/day). Patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of liraglutide or glimepiride. The analyses will be restricted to individuals with type 2 diabetes mellitus who have been previously treated with antidiabetic drugs. In the replication, previous anti-diabetic treatment was defined as the presence of at least 2 prescriptions for metformin within 6 months before and including cohort entry.
Sampling Method: Non-Probability Sample
Enrollment: 3474 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Relative Hazard of change in HbA1c from baseline to 26 weeks of treatment (end of follow-up) | 26-week follow-up window with a median follow-up time of 99 [84, 148] days
  Claims-based algorithm: relative hazard of change in HbA1c from baseline to 26 weeks of treatment (end of follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT05162183/Prot_SAP_000.pdf